CLINICAL TRIAL: NCT04694534
Title: e-SEP Cognition: Effectiveness of a Remediation Program Via a "Serious Game" on the Cognitive Functions of Multiple Sclerosis Patients: Controlled, Randomized, Multicentric Trial
Brief Title: Remediation Program Via a "Serious Game" for the Cognitive Functions of Multiple Sclerosis Patients
Acronym: E-SEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RC-P0066
Record Dates: First submitted 2020-12-16; First posted 2021-01-05 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis; Memory; Learning
Keywords: Multiple sclerosis; Serious game; Episodic memory learning capacities; Information processing speed capacities
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: 1 Control group
  1 Experimental group
Who Masked: Outcomes Assessor
Masking Description: This is a blinded study for neuropsychological assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remediation program via a "serious game" (Experimental): Classic care (recommended by the French Haute Autorité de Santé) accompanied by cognitive remediation by "serious game"
  Interventions: Diagnostic Test: Serious game
- Classic care (French Haute Autorité de Santé) (Placebo Comparator): Classic care (recommended by French Haute Autorité de Santé)
  Interventions: Diagnostic Test: Usual HAS care

INTERVENTIONS:
Diagnostic Test: Serious game — The serious game is accessible via an online platform, on a tablet: 4 20-minutes activities sessions per week must be carried out.
  The program format in the serious game form makes possible to simultaneously understand a large number of cognitive functions.
  Arms: Remediation program via a "serious game"
Diagnostic Test: Usual HAS care — The control group patients will follow the care they need, according to the HAS recommendations. Non-specific cognitive activities notebooks will be provided to them. They will be instructed to perform the 4 20-minutes sessions per week for 4 months.
  Arms: Classic care (French Haute Autorité de Santé)

SUMMARY:
The main goal of this study is to assess the effectiveness of a cognitive remediation program based on a "serious game" on the information processing speed evolution and the process of learning via episodic memory in multiple sclerosis patients.

DETAILED DESCRIPTION:
Cognitive impairment affects 40 to 70% multiple sclerosis patients. This condition is characterized by slower information processing, associated with deficits in episodic memory, attention and executive functions. These disorders appear early, regardless of functional impairment, in "benign" forms and in clinically isolated syndromes of multiple sclerosis. These disruptions can have a significant impact in the socio-professional and personal life of patients and also in the quality of life (job loss risks, daily activities limitations).

Even if these disorders are now well documented, remediation strategies remain less studied. Some studies show that the "training" methods, often used, do not seem suitable for clinical monitoring, with benefits that do not persist over time. Despite their impact on daily life, no specific care for planning abilities, mental inhibition and flexibility, or even social cognition, have been well studied until today. The same is true concerning metacognitive abilities. Finally, remedial techniques are time consuming and difficult to adapt to patients still in professional activity.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting or progressive multiple sclerosis people defined according to Mc Donald's criteria revised in 2005
* Age between ≥ 18 and ≤ 65 years old
* Cognitive complaint, with at least one deficient score at the initial neuropsychological examination (<5th percentile of the reference group), one of the scores of which concerns at least one BICAMS test
* Have not had a definite relapse for at least 6 weeks
* Be at least 4 weeks away from a corticosteroid bolus
* Lack of neuroleptic treatment
* Patient with an Internet connection
* Signed informed consent

Exclusion Criteria:

* Severe cognitive deficit defined by obtaining a deficit score in more than six cognitive processes at the initial neuropsychological assessment.
* Neuropsychological care
* Inability to receive oral and written information
* Inability to use the software (due in particular to motor and / or sensory difficulties),
* Neurological or psychiatric comorbidity, other than MS and anxiodepressive syndrome
* Patient with severe anxiodepressive syndrome (BDI> 27)
* Participation in an interventional study on cognitive functions
* Patient under legal protection, guardianship or curatorship
* Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-10-08 (Actual); Primary Completion 2026-04-04 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in the California Verbal Learning Test (CVLT) | Change from baseline at 4 and 10 months
  The California Verbal Learning Test (CVLT) begins with the examiner reading a list of 16 words. Patients listen to the list and report as many of the items as possible.
Change in the Brief Visuo-spatial Memory Test (BVMT) | Change from baseline at 4 and 10 months
  In the Brief Visuospatial/lMemory Test six abstract designs are presented for 10 sec. The display is removed from view and patients render the stimuli via pencil on paper manual responses. Each design receives from 0 to 2 points representing accuracy and location. Thus, scores range from 0 to 12.
Change in the Symbol Digit Modalities Test (SDMT) | Change from baseline at 4 and 10 months
  The Symbol Digit Modalities Test (SDMT) presents a series of nine symbols, each paired with a single digit in a key at the top of a standard sheet of paper. Patients are asked to voice the digit associated with each symbol as rapidly as possible for 90 sec. There is a single outcome measure: the number correct.

SECONDARY OUTCOMES:
Change in the Auditory-verbal spans in direct or reverse order | Change from baseline at 4 and 10 months
  This assessment is required to evaluate short time memory and working memory.
Change in the Stroop Color-Word Test | Change from baseline at 4 and 10 months
  This assessment is required to evaluate inhibition capacities and sensitivity to interference.
Change in the Trail Making Test | Change from baseline at 4 and 10 months
  This assessment is required to evaluate cognitive flexibility abilities.
Change in the Categorical and phonemic verbal fluency test | Change from baseline at 4 and 10 months
  This test is required to evaluate the spontaneous flexibility abilities.
Change in the Tower of London test | Change from baseline at 4 and 10 months
  This test is required to assess planning capacities.
Change in the Commission test | Change from baseline at 4 and 10 months
  This test assesses planning skills in a greener context than the Tower of London test.
Change in the Concentrated Attention Test | Change from baseline at 4 and 10 months
  This assessment is required to evaluate selective attention.
Change in the Paced Auditory Serial Addition Task (PASAT) | Change from baseline at 4 and 10 months
  This assessment is required to evaluate information processing speed and sustained attention.
Change in the Mac Nair Scale | Change from baseline at 4 and 10 months
  This self-evaluation is required to assess cognitive complaint. It is a 39-items questionnaire corresponding to symptoms. Every symptom is noted on an ordinal scale in 5 steps.It is a scale with 5 degrees of severity measuring the frequency of disorders as follows: 4 = very often, 3 = often, 2 = sometimes, 1 = rarely, 0 = never.
Change in the IPA (Participation and Autonomy Impact) Form | Change from baseline at 4 and 10 months
  This test is focused on the subject social participation and autonomy. is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. The standard cut-off scores are as follows:
  0-9: indicates minimal depression 10-18: indicates mild depression 19-29: indicates moderate depression 30-63: indicates severe depression.
Change in the BDI-II Scale (Beck Depression Inventory II) | Change from baseline at 4 and 10 months
  This scale is required to assess participants depressive orders. This is a 21-items self-questionnaire. Every item is rated from 0 (no problem) to 3 (maximum symptom severity). The depressive syndrome severity total score presents 4 intensity levels : 0-11 (no depression), 12-19 (mild depression), 20-27 (medium depression), 27 (severe depression).
Change in the State-Trait Anxiety Inventory (STAI Y) | Change from baseline at 4 and 10 months
  This scale is used to evaluate the participants level anxiety. It is a 20-items questionnaire. The patients identifie the frequency with which they usually feel the symptoms listed on a four-point Likert-type scale variant from 1: "never" on the 1 point side to 4: "always" on the 4 point side.
  The overall score varies between 20 and 80.
Change in the Visual Analogue Scale for Fatigue | Change from baseline at 4 and 10 months
  This scale allows patients to assess their fatigue. The patients locate their fatigue intensity on a 100-millimeters horizontal line.Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Change in the Apparent validity | Change from baseline at 4 and 10 months
  Face validity is based on a subjective assessment of the instrument's validity to assess the patient's attitude towards the tool, its degree of involvement and its acceptability.
Change in the EDSS score (Expanded disability status scale) | Change from baseline at 4 and 10 months
  This score is required to assess the patients functional and neurological level disability. This scale stretchs from 0 (no complaint and normal examen) to 10 (death caused by MS). The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist.
Frequency of game play per Week (in days) | Observance at 4 months
  This outcome is required to evaluate the instructions observance and play practices.
Game session lenght | Observance at 4 months
  This outcome is required to evaluate the instructions observance and play practices.
Time spent gaming | Observance at 4 months
  This outcome is required to evaluate the instructions observance and play practices.
Game performance : tests number per exercise | Observance at 4 months
  This outcome is required to evaluate the instructions observance and play practices. The performance will be evaluated by the tests number per exercise.
Game performance : difficulty levels | Observance at 4 months
  This outcome is required to evaluate the instructions observance and play practices. The performance will be evaluated by the difficulty levels.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Lenne, Principal Investigator — Hôpital Saint-Vincent de Paul
Locations (6):
- France (6):
  - CH Arras, Arras, Hauts-de-France
  - CH LENS, Lens, Hauts-de-France
  - CHRU, Lille, Hauts-de-France
  - Saint Vincent hospital, Lille, Hauts-de-France
  - Saint-Philibert hospital, Lomme, Nord
  - Charles Nicolle Hospital, Rouen, Normandy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lenne B, Degraeve B, Davroux J, Norberciak L, Kwiatkowski A, Donze C. Improving cognition in people with multiple sclerosis: study protocol for a multiarm, randomised, blinded trial of multidomain cognitive rehabilitation using a video-serious game (E-SEP cognition). BMJ Neurol Open. 2023 Nov 27;5(2):e000488. doi: 10.1136/bmjno-2023-000488. eCollection 2023. PMID 38033375